CLINICAL TRIAL: NCT07088133
Title: Clinical Trials of the Hepatitis B Sandwich Combination Therapy for Treating Patients Infected With Hepatitis B Virus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-250R2
Record Dates: First submitted 2025-07-05; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: HBV Infection; HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NA(s)+HT-102+FD-001 (Experimental)
  Interventions: Drug: NA(s)+HT-102+FD-001

INTERVENTIONS:
Drug: NA(s)+HT-102+FD-001 — Nucleos(t)ide analogues will be administrated throughout the entire treatment course; Patients will be injected with HT-102 once in Day1 (Week1), Day8 (Week2), Day15 (Week3), Day22 (Week4); Patients will be injected with FD-001 once in Day29 (Week5), Day57 (Week9), Day85 (Week13), Day113 (Week17), Day141 (Week21), Day169 (Week25) after confirmed reduction of serum HBsAg to below 10 IU/mL.

SUMMARY:
* Primary objective: The main objective of this study is to assess the efficacy and safety of a sandwich combination therapy in patients who were infected with HBV or have undergone surgery for hepatitis B virus (HBV)-related hepatocellular carcinoma (HCC). The primary efficacy endpoints are HBsAg seroconversion rate (HBsAg disappearance and HBsAb appearance), and HCC recurrence rate at week 49. Secondary Objective: To evaluate the safety of the HBV sandwich combination therapy through various safety indicators. Safety Indicators as follows: 1) Vital Signs: Monitoring systolic and diastolic blood pressure, pulse, respiration, and body temperature; 2) Physical Examination: Comprehensive physical assessments during the study; 3) 12-lead Electrocardiogram: Conducted to monitor cardiac health; 4) Clinical Laboratory Tests: Including blood routine, urine routine, blood biochemistry (focusing on liver and kidney function), coagulation function; 5) Injection Site Reactions: Monitoring for any local adverse effects from injections; 6) Adverse Events (AEs) and Serious Adverse Events (SAEs): Documentation of any AEs or SAEs occurring during treatment.
* Study Design: This study comprises three distinct stages:

  1. Screening Period (Weeks -4 to -1): 1) Informed consent will be obtained from participants; 2) Collect baseline data and perform various assessments which include: a) 12-lead ECG; b) Infectious disease screening; c) Blood biochemistry, routine blood, urine routine, coagulation function; d) Blood pregnancy test (for female subjects); e) Hepatitis B virus and serology examination; f) Antinuclear antibody testing; g) Imaging examinations.
  2. Treatment Period (Weeks 1 to 25): 1) Patients will receive ongoing nucleoside analogue treatment (NAs) throughout this stage; 2) Administer subcutaneous injections of the HBV monoclonal antibody HT-102 weekly for a total of 4 weeks (300 mg each time); 3) After treatment with HT-102, HBV serological and virological assessments will occur; 4) If serum HBsAg is below 10 IU/mL, proceed with therapeutic hepatitis B vaccine FD-001 (60 µg each time) every 4 weeks for a total of 6 doses; 5) If HBsAg is not below 10 IU/mL post HT-102, participants will enter the follow-up period directly.
  3. Follow-up Phase (Weeks 25 to 49): 1) Continue with original nucleoside analogue treatment for HBV; 2) Conduct follow-up visits every 12 weeks; 3) Each visit will involve recording vital signs, conducting physical examinations, ECG, laboratory tests (as noted in safety indicators), and testing for HBV and immunological parameters.
* End of Study:

The study concludes once the follow-up of the last enrolled subject is completed, analyzing the collected data to evaluate efficacy and safety endpoints.

- Note: Careful monitoring and adherence to protocols will be maintained to ensure participant safety and integrity of study data.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 weeks and ≤70 years, with an expected survival time of more than 12 months;
2. HCC subjects who have undergone radical surgery or ablation therapy, and no residual tumor lesions in the liver (R0 resection) were found in the postoperative review, and the postoperative pathological specimens confirmed that they were primary liver cancer and had evidence of chronic hepatitis, no evidence of extrahepatic metastasis, and did not require postoperative adjuvant therapy for low- and medium-risk subjects;
3. Barcelona Clinic Liver Cancer (BCLC) stage 0 or A; Child-Pugh liver function grade A during the screening period, ECOG score 0;
4. No imaging evidence of invasion of the main portal vein branches; Clinically diagnosed with chronic hepatitis B (serum HBsAg positive ≥6 months);
5. Understand and are willing to sign the informed consent form, and are willing to comply with all research procedures specified in this study;
6. Females of childbearing age have negative blood pregnancy tests, and subjects of childbearing age (including male subjects) have no pregnancy plans in the next 3 months and voluntarily take effective contraceptive measures;
7. Have received antiviral treatment with nucleoside (acid) analogs such as tenofovir alafenamide fumarate (TAF), tenofovir disoproxil fumarate (TDF) or entecavir (ETV) for at least one year, and have received stable treatment with nucleoside (acid) analogs for ≥2 months during the screening period, and agree to continue using them during the study. For subjects who have previously used non-first-line nucleoside (acid) analogs such as lamivudine/adefovir/telbivudine, they agree to switch to first-line ETV/TAF/TDF/TMF and continue to use;
8. HBV DNA <2000 copies/ml or 200 IU/ml at screening; HBsAg >10IU/ml and <3000 IU/ml;
9. With adequate organ and bone marrow function, laboratory test values meet the following requirements:

   1. Routine blood test: absolute neutrophil count (ANC) ≥1.5×109 /L; platelet count (PLT) ≥90×109 /L; hemoglobin content (HGB) ≥90g/L;
   2. Liver function: serum albumin >35g/L; serum total bilirubin (TBIL) ≤2.5×upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤10.0×ULN; alkaline phosphatase (ALP) ≤2.5×ULN;
   3. Coagulation function: international normalized ratio (INR), prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN. If the subject is taking anticoagulant therapy such as warfarin or heparin, it is necessary to ensure that the protocol requirements are met when the drug is stopped or not used;
   4. Urinalysis: urine protein negative or 24-hour urine protein quantitative ≤ ULN. Screening urine protein 1+ can be further confirmed by rechecking urine routine, and 24-hour urine protein quantitative test can be performed if necessary;
   5. Electrolytes are normal or normal after treatment or are judged by the researcher to be abnormal and have no clinical significance;
   6. Creatinine clearance (Ccr) >50 mL/(min·1.73m2)

Exclusion Criteria:

1. Liver transplant or liver transplant candidate; previous or current diagnosis of psychiatric illness or major depression;
2. Other malignancies, except for carcinoma in situ of the cervix and/or non-melanoma skin cancer and superficial bladder tumors (Ta [non-invasive tumor], Tis [breast cancer in situ], and T1 [tumor invading the lamina propria]). Any cancer that has been effectively treated for more than 3 years before participating in the study is allowed;
3. Those with clinical symptoms of brain metastases, or other evidence that the subjects' brain metastases have not been controlled, and/or meningeal metastases, are judged by the researchers to be unsuitable for inclusion;
4. Past or current ascites, esophageal or gastric varicose bleeding caused by portal hypertension, hepatorenal syndrome, hepatic encephalopathy or liver failure, suspected cirrhosis or compensated cirrhosis, etc.;
5. Liver diseases caused by other reasons, including chronic alcoholic hepatitis, drug-induced hepatitis, autoimmune hepatitis, hepatolenticular degeneration and hemochromatosis;
6. Interferon or pegylated interferon treatment or other strong immunomodulators such as adrenocortical hormone, thymosin a1, thymosin 5 peptide, etc. were used within 12 weeks before the first use of the study drug, or interferon or pegylated interferon treatment or other strong immunomodulators such as adrenocortical hormone, thymosin a1, thymosin 5 peptide, etc. are planned to be used during the trial;
7. Immunosuppressants used within 6 months before the first use of the study drug; corticosteroids used for 1 week or more within 6 months before the first use of the study drug (except topical or inhaled corticosteroids);
8. Positive hepatitis C virus (HCV), hepatitis D virus (HDV), Treponema pallidum (TP) antibodies or human immunodeficiency virus (HIV) antibodies;
9. A history of clinically significant cardiovascular disease, including but not limited to: myocardial infarction, uncontrolled angina pectoris, viral myocarditis, stroke or other grade 3 or above cardiovascular and cerebrovascular events within 6 months before the first administration of this study drug; any supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention, left ventricular ejection fraction (LVEF) <50%, congestive heart failure of New York Heart Association (NYHA) heart function class III or IV, uncontrolled hypertension [systolic blood pressure (SBP) ≥160mmHg and/or diastolic blood pressure (DBP) ≥100mmHg after standard treatment or history of hypertensive crisis or hypertensive encephalopathy];
10. Any life-threatening bleeding event in the past 3 months, including the need for transfusion, surgery or local treatment, and continuous drug treatment;
11. Those who are known or may be allergic to HT-102 or FD-001 and its excipients; those who have a known history of allergy to hepatitis B vaccination;
12. Participated in another clinical trial of a study drug or biological agent within 30 days or 5 half-lives before the first use of the study drug;
13. Pregnant or breastfeeding women; those who the investigator believes are not suitable for participation in this trial due to other reasons;
14. Active autoimmune diseases Patients with active autoimmune diseases or known history of autoimmune diseases who require systemic hormone or immunosuppressant treatment, including but not limited to rheumatoid arthritis, systemic lupus erythematosus, Wegener's granulomatosis, Sjögren's syndrome, inflammatory bowel disease, multiple sclerosis, myasthenia gravis, myositis, autoimmune hepatitis, vasculitis, immune thrombocytopenic purpura, autoimmune hemolytic anemia and glomerulonephritis. Excluded: Subjects with endocrine diseases that can be controlled by HRT (such as hypothyroidism, type 1 diabetes, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Positive convention rate of HBsAb | through study completion, an average of 49 weeks
  evaluate the seroconversion rate of HBsAg (defined as the loss of HBsAg with the concurrent appearance of anti-HBs antibodies).

SECONDARY OUTCOMES:
Proportion of subjects with ≥ 0.5 log or ≥1 log reduction in serum HBsAg levels from baseline | week4, 13, 25, 37 and 49 after administraton
  to evaluate the efficacy of NA(s)+HT-102+FD-001
HBsAg changes | week4, 13, 25, 37 and 49 after administraton.
  to evaluate the efficacy of NA(s)+HT-102+FD-001
HBsAg clearance rate | week4, 13, 25 and 37 after administraton.
  HBsAg clearance rate defined as undetectable HBsAg or HBsAg below 10 IU/mL
HBsAg seroconversion rate | week4, 13, 25, 37 and 49 after administration
  HBsAg seroconversion rate defined as loss of HBsAg with concurrent development of HBsAb
HBeAg seroconversion rate | week4, 13, 25, 37 and 49 after administration
  HBeAg seroconversion rate defined as disappearance of HBeAg with concurrent appearance of HBeAb
HBeAg clearance rate | weeks 4, 13, 25, 37 and 49
  HBeAg clearance rate defined as undetectable HBeAg or HBeAg below 10 IU/mL
Time from initiation of HT-102 administration to achievement of HBsAg clearance | through study completion, an average of 49 weeks
  to evaluate the efficacy of NA(s)+HT-102+FD-001
Time from initiation of HT-102 administration to achievement of HBsAg seroconversion. | through study completion, an average of 49 weeks
  to evaluate the efficacy of NA(s)+HT-102+FD-001
HBsAb change | week4, 13, 25, 37 and 49 after administration
  to evaluate the efficacy of NA(s)+HT-102+FD-001
Changes from baseline in other HBV-related biomarkers including HBV DNA, HBeAg, anti-HBe (HBeAb), HBcAg, anti-HBc (HBcAb), and liver function parameters (ALT and AST). | week4, 13, 25, 37 and 49 after administration
  to evaluate the efficacy of NA(s)+HT-102+FD-001